CLINICAL TRIAL: NCT04122781
Title: Treatment of Pediatric Supracondylar Humeral Fractures With Novel Kirschner Wire Fixation Devices: A Prospective Comparative Study
Brief Title: Treatment of Pediatric Supracondylar Humeral Fractures With Novel Kirschner Wire Fixation Devices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRPD1J1171
Record Dates: First submitted 2019-09-22; First posted 2019-10-10 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2019-09

CONDITIONS: Supracondylar Humerus Fracture
Keywords: supracondylar humerus fracture; Kirschner wire

STUDY DESIGN:
Intervention Model Description: A prospective Comparative Study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with novel K-wire fixation devices (Experimental): Patients with supracondylar humeral fractures treated by percutaneous K-wire fixation and novel K-wire fixation devices
  Interventions: Device: Novel K-wire fixation devices
- without novel K-wire fixation devices (Active Comparator): Patients with supracondylar humeral fractures treated by percutaneous K-wire fixation
  Interventions: Device: Novel K-wire fixation devices

INTERVENTIONS:
Device: Novel K-wire fixation devices — The patients received surgery using novel K-wire fixation devices

SUMMARY:
A novel K-wire external fixation device was developed by the investigators. The K-wires can be connected by the device. After connection, the structure of the K-wires is transformed to an external skeletal fixator. Therefore, the K-wires are stabilized and unable to migrate independently. The stability of fracture fixation is better in patient with this K-wire external fixation device.

The purposes of this study are to optimize the K-wire external fixation device and test its function in real clinical practice.

DETAILED DESCRIPTION:
Supracondylar humeral fractures are the most common elbow fractures in children. Closed reduction and internal fixation using percutaneous Kirschner wires (K-wires) are widely recommended for Gartland type II and III fractures. After percutaneous pinning, the K-wires are bent at the skin edge and cut. The cutoff point is about 1 cm outside of the skin.

The diameters of the K-wires are between 1.5-3.0 mm. The surface of the K-wire is smooth. Therefore, the K-wires are easy to rotation and migration. Proximal migration or rotation of a K-wire could injure the skin. Distal migration of a K-wire could result in loss of reduction and fixation. Therefore, stabilization of the K-wires is important.

A novel K-wire external fixation device was developed by the investigators. The K-wires can be connected by the device. After connection, the structure of the K-wires is transformed to an external skeletal fixator. Therefore, the K-wires are stabilized and unable to migrate independently. The stability of fracture fixation is better in patient with this K-wire external fixation device.

The investigators got a one-year grant from the Ministry of Science and Technology in Taiwan last year. The preliminary data revealed that the torque and torsional stiffness with the K-wire external fixation device was greater than traditional pinning.

The purposes of this study are to optimize the K-wire external fixation device and test its function in real clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric supracondylar humeral fracture
* Patients receiving closed reduction and percutaneous pinning

Exclusion Criteria:

* Open fracture
* Open reduction
* Neurovascular exploration

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Radiographs measurement | through study completion, an average of 1 year
  Baumann angle and the location of anterior humeral line on the radiographs
Elbow range of motion | through study completion, an average of 1 year
  Elbow flexion an extension angle
Pin sites condition | 4 weeks
  The pin sites were inspected and graded according to the system of Dahl. Grade 0 was normal skin, grade 1 was pain or erythema without discharge, grade 2 was serous discharge, grade 3 was purulent discharge, grade 4 was radiographic osteolysis and grade 5 was ring sequestrum or osteomyelitis.

CONTACTS AND LOCATIONS:
Overall Officials: Hsuan-Kai Kao, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No